CLINICAL TRIAL: NCT03486197
Title: Phase II Trial of Neutron Radiotherapy With Concurrent Checkpoint Inhibitor Immunotherapy (Pembrolizumab) in Patients With Advanced Urothelial Carcinoma
Brief Title: Neutron Radiation Therapy and Pembrolizumab in Treating Participants With Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jing Zeng, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9940; NCI-2018-00412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9940 (Other: Fred Hutch/University of Washington Cancer Consortium); RG3118000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Pembrolizumab, neutron radiation therapy) (Experimental): Participants receive pembrolizumab IV on days 1 and 22. On day 23, participants may undergo an optional tumor biopsy and receive 3-5 treatments of neutron radiation therapy over 2 weeks on days 23-42. Participants receive pembrolizumab IV on day 43 and continue per standard of care in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo neutron radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well neutron radiation therapy and pembrolizumab work in treating participants with urothelial carcinoma that has spread to other places in the body. Neutron radiation therapy uses high energy neutrons to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving radiation therapy and pembrolizumab may work better than radiation alone in treating participants with urothelial carcinoma that has spread to other places in the body.

DETAILED DESCRIPTION:
OUTLINE:

Participants receive pembrolizumab intravenously (IV) on days 1 and 22. On day 23, participants may undergo an optional tumor biopsy and receive 3-5 treatments of neutron radiation therapy over 2 weeks on days 23-42. Participants receive pembrolizumab IV on day 43 and continue per standard of care in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of urothelial carcinoma
* At least two sites of disease that are measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Eligible for checkpoint inhibitor immunotherapy (pembrolizumab) per standard of care
* No history of autoimmune disease requiring systemic therapy (e.g. steroids or biologic agents)
* Absolute neutrophil count (ANC) ≥ 1500 /mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin > 9 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR ≥ 60 mL/min
* Total bilirubin ≤ 1.5 ULN OR direct bilirubin ≤ ULN if total bilirubin > 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN OR < 5 x ULN if patient has liver metastasis
* Albumin >= 2.5 g/dL
* International normalized ratio (INR) or PT ≤ 1.5 x ULN unless on anticoagulation therapy, in which case prothrombin time (PT) or partial thromboplastin time (PTT) should be in the therapeutic range
* PTT ≤ 1.5 x ULN unless on anticoagulation therapy, in which case PT or PTT should be in the therapeutic range
* Eligible for neutron radiation treatment to 1-3 sites of metastatic disease (lesions do not have to be symptomatic)
* No steroids for at least 2 weeks prior to enrollment, and patient must not be expected to require steroids during the study period
* Zubrod performance status 0-2
* Patient must sign study specific informed consent prior to study entry
* Patients who are sexually active must use medically acceptable forms of contraception
* Life expectancy must be > 3 months

Exclusion Criteria:

* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a known additional malignancy that is progressing or requires active treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has received a live vaccine within 30 days of planned start of study therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided there is no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Seattle, WA
  participants
    United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Per Immune-modified Response Evaluation Criteria in Solid Tumors
Description: Overall response rate will be calculated as the percentage of patients achieving a partial response or complete response.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
Number analyzed (Participants) | 12
Participants | 6

2. Secondary Outcome: Overall Survival
Description: Final statistical analyses of OS will consist of Kaplan-Meier estimation.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
Number analyzed (Participants) | 12
percentage of participants | 62 [51 to 74]

3. Secondary Outcome: Progression-free Survival
Description: Final statistical analyses of PFS will consist of Kaplan-Meier estimation.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
Number analyzed (Participants) | 12
percentage of participants | 55 [41 to 68]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during radiation treatment weekly during physician visits, and during each pembrolizumab infusion with a physician visit for up to 1 year.
Description: CTCAE v4 was used to grade adverse events for up to 1 months after study enrollment.
Arm/Group | Treatment (Pembrolizumab, Neutron Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 6/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Neutron Radiation Therapy) (N=12)
Myositis Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Kidney Injury Grade 3 (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Neutron Radiation Therapy) (N=12)
Fatigue Grade 2 (General disorders) | 5 (5)
Gastritis Grade 2 (Gastrointestinal disorders) | 2 (2)
Pancreatitis Grade 2 (Gastrointestinal disorders) | 1 (1)
Acute Kidney Injury Grade 2 (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03486197/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03486197/ICF_002.pdf